CLINICAL TRIAL: NCT07364162
Title: Exogenous Ketone Ester Supplementation in ICU Delirium (KETONES ICU)
Brief Title: Exogenous Ketone Supplementation in ICU Delirium
Acronym: KETONES-ICU
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Smith, Pulmonary & Critical Care Medicine Fellow, Vanderbilt University Medical Center, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U16370
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: ICU Delirium; Critical Illness
Keywords: ICU; Intensive Care Unit; Critical care; Critical illness; Ketones
MeSH Terms: conditions — Critical Illness; Ketosis | interventions — (R)-3-hydroxybutyl (R)-3-hydroxybutyrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketone supplement (Experimental)
  Interventions: Drug: Ketone supplementation
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketone supplementation — Ketone monoester diluted to a total volume of 74 mL with water and administered enterally (oral/feeding tube). Dosing is protocolized with an initial dose of 25 g and subsequent dose titration based on serum β-hydroxybutyrate levels to target a prespecified serum β-hydroxybutyrate range, administered every 6 hours for up to 7 days (or ICU discharge or death, whichever occurs first).
  Other Names: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate; D-β-hydroxybutyrate monoester; D-BHB monoester; ketone monoester; (R)-hydroxybutyl (R)-3-hydroxybutyrate;; [(3R)-3-hydroxybutyl] (3R)-3-hydroxybutanoate)
  Arms: Ketone supplement
Drug: Placebo — Placebo consists of 74 mL of dextrose 50% in water (D50W) plus 50 mg sucrose octaacetate for taste matching; administered enterally (oral/feeding tube) on the same schedule as the experimental arm.
  Arms: Placebo

SUMMARY:
Delirium is a common syndrome in intensive care unit (ICU) patients. Those experiencing delirium may suddenly feel confused, have trouble thinking clearly, struggle to pay attention, or see and hear things that are not real. Delirium is associated with worse long-term outcomes such as cognitive impairment, depression, and PTSD (post-traumatic stress disorder). This study examines whether an investigational medical-grade ketone supplement drink (ketone monoester [brand name: Ultrapure Ketone Monoester]) is safe and feasible to use in ICU patients, and to look for signals that it might reduce delirium or shorten its duration compared to a volume-, taste-, and calorie-matched placebo.

DETAILED DESCRIPTION:
Delirium is a prevalent neuropsychiatric syndrome characterized by an acute disturbance in attention, cognition, and consciousness. It is associated with significant morbidity, mortality, and healthcare expenditures. Recent research has provided evidence supporting the connection between brain metabolism and delirium. During states of increased systemic inflammation, such as sepsis or trauma, the brain experiences a mismatch between energy supply and demand, which is commonly associated with delirium, especially in those with preexisting cognitive impairment.

In critically ill patients, mitochondrial dysfunction occurs in the setting of systemic inflammation, contributing to increased blood-brain barrier permeability and neuroinflammation. The downstream consequence of this is microglial activation, which amplifies the inflammatory response through the release of pro-inflammatory cytokines. The resultant mitochondrial dysfunction leads to impaired oxidative phosphorylation, decreased adenosine triphosphate (ATP) production, and increased reactive oxygen species production. In response to systemic inflammation, microglia transition to a pro-inflammatory phenotype characterized by increased aerobic glycolysis. This metabolic reprogramming depletes glucose availability for neurons and exacerbates the cerebral energy deficit. Emerging evidence suggests that activated microglia compete with neurons for metabolic substrates during inflammation. Activated microglia exhibit metabolic flexibility, shifting toward increased glycolysis to meet their heightened energy and biosynthetic demands. This competition for nutrients exacerbates the neuronal energy deficit and increases metabolic stress. The investigators hypothesize that this brain energy deficit contributes to the cognitive and neurological symptoms characteristic of delirium.

Ketones, such as β-hydroxybutyrate, are the brain's secondary source of energy when glucose is not available. After transport across the blood-brain barrier, β-hydroxybutyrate is metabolized to acetyl-CoA (acetyl coenzyme A), thereby directly entering the tricarboxylic acid cycle, bypassing the glycolytic bottleneck, to produce ATP. In addition to serving as a substrate for ATP production, ketones support mitochondrial function, limit oxidative stress, and reduce neuroinflammation. Ketones confer a two-fold therapeutic advantage in the setting of nutrient competition. Not only do they support neuronal oxidative phosphorylation by bypassing impaired glycolysis, but they also promote anti-inflammatory microglial phenotypes, inhibit inflammasome activation, and support metabolic reprogramming. This dual effect further reduces microglial glucose demand, enhancing neuronal substrate availability.

The investigators propose a prospective, randomized, placebo-controlled pilot study of exogenous ketone ester supplement administration in 40 critically ill patients to assess the safety and feasibility of this novel intervention and to generate preliminary data on its efficacy in reducing ICU delirium, as measured by delirium and coma free days (DCFDs). Exogenous ketones have been shown to support brain energetics and reduce neuroinflammation, directly targeting pathways implicated in the development of delirium. By reducing the duration of delirium or preventing its onset, this research has the potential to improve long-term cognitive outcomes for ICU survivors. The investigators propose enrolling adult patients at the time of ICU admission, with randomization to either an enteral ketone ester treatment group or a taste, volume, and calorie-matched dextrose-containing placebo. The study drug or placebo will be administered at the time of enrollment, within 24 hours of ICU admission, and every six hours thereafter for up to 7 days until ICU discharge, or death, whichever occurs first. Ketone administration will be continued after the diagnosis of delirium. In accordance with prior studies, the initial dose of β-hydroxybutyrate will be 25 g; however, subsequent doses will be titrated to maintain serum β-hydroxybutyrate levels between 1.5 and 3.5 mM, with protocolized monitoring of vital signs, serum pH, glucose levels, and adverse gastrointestinal effects. Delirium will be assessed using the Confusion Assessment Method for the ICU (CAM-ICU) delirium screening tool twice daily for a period of 7 days.

This pilot study will assess the feasibility, safety, and tolerability of oral exogenous ketone supplementation in critically ill patients. The goal is to demonstrate that ketone administration is well-tolerated, with no significant safety concerns, consistent with prior evidence that oral ketones can be administered safely, even in vulnerable patient populations. Successful completion of this aim will establish a safety profile for ketone use in the ICU, which is essential before adopting this novel therapy for critically ill patients. The investigators hypothesize that patients receiving ketones will have more DCFDs compared to those receiving a placebo. The investigators will also perform an exploratory analysis of the biological impact of ketone therapy by examining biomarkers associated with delirium and ketone metabolism through serial measurement of serum levels of peripheral inflammatory mediators, metabolic stress assays, β-hydroxybutyrate levels, and markers of central nervous system (CNS) injury.

Ketones offer a promising novel therapeutic option for delirium. By targeting the underlying neurometabolic and neuroinflammatory changes associated with delirium, they support energy production, decrease oxidative stress, and modulate inflammation. Patients with preexisting cognitive impairment, such as those with mild cognitive impairment or Alzheimer's dementia, exhibit a baseline brain energy gap due to impaired cerebral glucose metabolism. This chronic energy deficit increases the vulnerability of the aging brain to delirium. Furthermore, the neurometabolic consequences of delirium in those with preexisting cognitive impairment exacerbate the brain energy gap, accelerating cognitive decline. The safety, tolerability, and rapid induction of ketosis following oral administration of ketone esters, in addition to the aforementioned beneficial effects, suggest this may be a therapy that could be initiated upon ICU admission as a potential preventative measure in those patients at risk. Ketones have the potential to transform delirium management and improve patient care; however, this clinical trial is required to evaluate the safety and efficacy of oral ketone ester supplementation in reducing the incidence, severity, and duration of delirium in critically ill patients.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients (≥18 years old) admitted to the medical intensive care unit.
2. Current ICU admission with anticipated ICU stay ≥24 hours.
3. Enteral access in place, planned enteral access placement, or PO intake appropriate, and the ability to receive enteral dosing within 24 hours of enrollment.
4. Ability to complete delirium assessments (CAM-ICU feasible) at time of enrollment.

Exclusion criteria:

1. Severe metabolic acidosis at enrollment: blood gas pH <7.20 or bicarbonate < 8 mmol/L.
2. Diabetic ketoacidosis as an ICU admission diagnosis or hyperketonemia from any ketoacidosis state.
3. Hypoglycemia as an ICU admission diagnosis or glucose <60 mg/dL.
4. Patients with a history of type 1 diabetes mellitus.
5. Hemoglobin <7.0.
6. Renal failure requiring dialysis initiated or anticipated at enrollment (CRRT or iHD).
7. Fulminant hepatic failure or AST/ALT > 5× ULN or total bilirubin > 3 mg/dL.
8. Refractory shock (defined as norepinephrine dose ≥20 µg/min or use of a second vasopressor agent).
9. Pregnancy (positive urine/serum hCG at screening or known pregnancy).
10. Uncontrolled ileus or gastrointestinal condition, such as an upper gastrointestinal bleed, preventing enteral dosing.
11. SGLT2 inhibitor use within the prior 7 days.
12. ADH/ALDH inhibitors (e.g., fomepizole, disulfiram) use in the prior 7 days or planned.
13. Severe dementia or neurodegenerative disease, defined as either impairment that prevents the patient from living independently at baseline or IQCODE >4.5, measured using a patient's qualified surrogate. This exclusion also pertains to mental illnesses requiring long-term institutionalization, acquired or congenital intellectual disability, severe neuromuscular disorders, Parkinson's disease, and Huntington's disease. It also excludes patients with severe deficits due to structural brain diseases such as stroke, intracranial hemorrhage, cranial trauma, malignancy, anoxic brain injury, or cerebral edema.
14. Benzodiazepine dependency or alcohol dependency based on the medical team's decision to institute a specific treatment plan involving benzodiazepines (either as continuous infusions or intermittent intravenous boluses) for this dependency.
15. Active seizures during this ICU admission being treated with intravenous benzodiazepines.
16. Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family/medical team (e.g., likely to withdraw life support measures within 24 hours of screening).
17. Admission to ICU only for post-operative monitoring or frequent neurologic assessments.
18. Incarcerated status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Proportion of participants achieving target peak serum β-hydroxybutyrate (1.5-3.5 mmol/L) on at least 50% of dosing days | From enrollment through study day 7 or ICU discharge.
  Peak serum β-hydroxybutyrate will be measured once daily using safety laboratories drawn 60-90 minutes after the morning ketone dose to capture the post-dose peak level. A dosing day will be considered successful if the measured peak serum β-hydroxybutyrate is within 1.5-3.5 mmol/L. The primary feasibility outcome is the proportion of participants in the ketone group who have successful peak serum β-hydroxybutyrate measurements on ≥50% of dosing days during the dosing period. Feasibility will be considered met if ≥70% of participants in the ketone group meet this criterion.
Safety and tolerability: Number of participants with ≥1 prespecified safety or tolerability event | From enrollment through study day 7.
  A prespecified safety or tolerability event is defined as any of the following occurring from enrollment through study day 7: acid-base abnormality (blood gas pH <7.20 or serum bicarbonate <8 mmol/L), off-target hyperketonemia (peak serum β-hydroxybutyrate >3.5 mmol/L despite dose reduction), hypoglycemia (<60 mg/dL), renal or hepatic safety signal (new dialysis initiation; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5× upper limit of normal, or total bilirubin >3 mg/dL without alternative explanation), hemodynamic instability temporally related to dosing, or gastrointestinal symptoms (nausea, vomiting, diarrhea, cramping) recorded as tolerability adverse events. The outcome will be summarized as the number of participants with ≥1 prespecified event by treatment arm.

SECONDARY OUTCOMES:
Feasibility: Proportion of scheduled post-dose serum β-hydroxybutyrate draws completed | From enrollment through study day 7 or ICU discharge.
  The proportion of scheduled daily post-dose serum β-hydroxybutyrate draws that are successfully collected during the dosing period will be calculated and summarized. Feasibility performance will be summarized relative to a target of ≥80% completion.
Feasibility: Proportion of post-dose serum β-hydroxybutyrate measurements >4.0 mmol/L | From enrollment through study day 7 or ICU discharge.
  Using the daily post-dose peak serum β-hydroxybutyrate measurements obtained during the dosing period, the proportion of measurements with β-hydroxybutyrate >4.0 mmol/L will be calculated and summarized by treatment arm. Performance will be summarized relative to a target of <10% of measurements >4.0 mmol/L.
Feasibility: Adherence to ketone dose-titration algorithm | From enrollment through study day 7 or ICU discharge.
  Adherence will be defined as the proportion of dosing decisions during the dosing period that follow the prespecified dose-titration algorithm based on post-dose serum β-hydroxybutyrate results and protocol-defined dose adjustment rules. Adherence will be summarized relative to a target of ≥80%.
Delirium- and coma-free days (DCFDs) through study day 7 | From enrollment through study day 7.
  Delirium- and coma-free days (DCFDs) is defined as the number of days from enrollment through study day 7 during which participants are alive and free of both delirium and coma. Delirium is defined as any positive assessment on the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) administered twice daily while participants remain in the intensive care unit. Coma is defined according to the study protocol. DCFDs will be summarized by treatment arm.
Delirium severity score on the Confusion Assessment Method for the Intensive Care Unit-7 (CAM-ICU-7) scale | From enrollment through study day 7.
  Delirium severity will be measured and reported using the Confusion Assessment Method for the Intensive Care Unit-7 (CAM-ICU-7) delirium severity scale. The CAM-ICU-7 score ranges from 0 (minimum) to 7 (maximum), with higher scores indicating worse (more severe) delirium. CAM-ICU-7 scores will be summarized by treatment arm over the assessment period.
Change from baseline in serum interleukin-1 beta (IL-1β) concentration | From enrollment through study day 7.
  Serum interleukin-1 beta (IL-1β) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum interleukin-6 (IL-6) concentration | From enrollment through study day 7.
  Serum interleukin-6 (IL-6) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum interleukin-8 (IL-8) concentration | From enrollment through study day 7.
  Serum interleukin-8 (IL-8) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum interleukin-10 (IL-10) concentration | From enrollment through study day 7.
  Serum interleukin-10 (IL-10) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum interleukin-18 (IL-18) concentration | From enrollment through study day 7.
  Serum interleukin-18 (IL-18) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum C-reactive protein (CRP) concentration | From enrollment through study day 7.
  Serum C-reactive protein (CRP) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum monocyte chemoattractant protein-1 (MCP-1) concentration | From enrollment through study day 7.
  Serum monocyte chemoattractant protein-1 (MCP-1) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum tumor necrosis factor alpha (TNF-α) concentration | From enrollment through study day 7.
  Serum tumor necrosis factor alpha (TNF-α) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Peak serum beta-hydroxybutyrate concentration following dosing | From enrollment through study day 7 or ICU discharge.
  Peak serum beta-hydroxybutyrate concentration will be measured once daily using a post-dose blood draw collected 60-90 minutes after the morning dose and reported in mmol/L by treatment arm.
Change from baseline in serum neurofilament light chain (NfL) concentration | From enrollment through study day 7.
  Serum neurofilament light chain (NfL) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum glial fibrillary acidic protein (GFAP) concentration | From enrollment through study day 7.
  Serum glial fibrillary acidic protein (GFAP) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.
Change from baseline in serum brain-derived neurotrophic factor (BDNF) concentration | From enrollment through study day 7.
  Serum brain-derived neurotrophic factor (BDNF) concentration will be measured at baseline and on study days 1, 3, 5, and 7 and reported as change from baseline by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: E. Wes Ely, MD, MPH, Study Director — Vanderbilt University Medical Center; Ryan J Smith, MD, JD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) for all randomized participants that underlie reported results, including: baseline demographics and clinical characteristics; eligibility variables; treatment assignment and dosing history; serum β-hydroxybutyrate and other protocol safety labs (e.g., glucose, acid-base measures); delirium/coma assessments (CAM-ICU, CAM-ICU-7) and derived delirium- and coma-free days through study day 7; key clinical outcomes (e.g., ICU/hospital length of stay, mortality); adverse events, dose holds/reductions/discontinuations; and research biomarker assay results. A data dictionary will be provided. Direct identifiers and free-text clinical notes will not be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 9 months after publication of the primary results and will remain available for 36 months following publication.
Access Criteria: De-identified IPD and supporting documents will be shared with qualified researchers who submit a methodologically sound proposal. Access requires approval by the study team, execution of a data use agreement, and IRB/ethics approval as applicable. Data will be provided via secure electronic transfer. Requestors must agree not to attempt re-identification and to use the data only for the approved purpose.

REFERENCES:
- [Background] Smith R, Harrison F, Bastarache J, Williams Roberson S, Zaganjor E, Pandharipande P, Rice T, Ely W. Potential therapeutic benefit of exogenous ketone ester administration in delirium: a narrative review. Crit Care. 2025 Oct 7;29(1):424. doi: 10.1186/s13054-025-05680-5. PMID 41057929
- [Background] Girard TD, Exline MC, Carson SS, Hough CL, Rock P, Gong MN, Douglas IS, Malhotra A, Owens RL, Feinstein DJ, Khan B, Pisani MA, Hyzy RC, Schmidt GA, Schweickert WD, Hite RD, Bowton DL, Masica AL, Thompson JL, Chandrasekhar R, Pun BT, Strength C, Boehm LM, Jackson JC, Pandharipande PP, Brummel NE, Hughes CG, Patel MB, Stollings JL, Bernard GR, Dittus RS, Ely EW; MIND-USA Investigators. Haloperidol and Ziprasidone for Treatment of Delirium in Critical Illness. N Engl J Med. 2018 Dec 27;379(26):2506-2516. doi: 10.1056/NEJMoa1808217. Epub 2018 Oct 22. PMID 30346242
- [Background] Saris CGJ, Timmers S. Ketogenic diets and Ketone suplementation: A strategy for therapeutic intervention. Front Nutr. 2022 Nov 15;9:947567. doi: 10.3389/fnut.2022.947567. eCollection 2022. PMID 36458166
- [Background] Hou L, Yang J, Li S, Huang R, Zhang D, Zhao J, Wang Q. Glibenclamide attenuates 2,5-hexanedione-induced neurotoxicity in the spinal cord of rats through mitigation of NLRP3 inflammasome activation, neuroinflammation and oxidative stress. Toxicol Lett. 2020 Oct 1;331:152-158. doi: 10.1016/j.toxlet.2020.06.002. Epub 2020 Jun 6. PMID 32522579
- [Background] Oh U, Woolbright E, Lehner-Gulotta D, Coleman R, Conaway M, Goldman MD, Brenton JN. Serum neurofilament light chain in relapsing multiple sclerosis patients on a ketogenic diet. Mult Scler Relat Disord. 2023 May;73:104670. doi: 10.1016/j.msard.2023.104670. Epub 2023 Mar 25. PMID 36996634
- [Background] Bock M, Steffen F, Zipp F, Bittner S. Impact of Dietary Intervention on Serum Neurofilament Light Chain in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2021 Nov 11;9(1):e1102. doi: 10.1212/NXI.0000000000001102. Print 2022 Jan. PMID 34764215
- [Background] McDougall A, Bayley M, Munce SE. The ketogenic diet as a treatment for traumatic brain injury: a scoping review. Brain Inj. 2018;32(4):416-422. doi: 10.1080/02699052.2018.1429025. Epub 2018 Jan 23. PMID 29359959
- [Background] Youm YH, Nguyen KY, Grant RW, Goldberg EL, Bodogai M, Kim D, D'Agostino D, Planavsky N, Lupfer C, Kanneganti TD, Kang S, Horvath TL, Fahmy TM, Crawford PA, Biragyn A, Alnemri E, Dixit VD. The ketone metabolite beta-hydroxybutyrate blocks NLRP3 inflammasome-mediated inflammatory disease. Nat Med. 2015 Mar;21(3):263-9. doi: 10.1038/nm.3804. Epub 2015 Feb 16. PMID 25686106
- [Background] Prins M, Greco T, Alexander D, Giza CC. The pathophysiology of traumatic brain injury at a glance. Dis Model Mech. 2013 Nov;6(6):1307-15. doi: 10.1242/dmm.011585. Epub 2013 Sep 12. PMID 24046353
- [Background] Xu Q, Zhang Y, Zhang X, Liu L, Zhou B, Mo R, Li Y, Li H, Li F, Tao Y, Liu Y, Xue C. Medium-chain triglycerides improved cognition and lipid metabolomics in mild to moderate Alzheimer's disease patients with APOE4-/-: A double-blind, randomized, placebo-controlled crossover trial. Clin Nutr. 2020 Jul;39(7):2092-2105. doi: 10.1016/j.clnu.2019.10.017. Epub 2019 Oct 22. PMID 31694759
- [Background] Ota M, Matsuo J, Ishida I, Takano H, Yokoi Y, Hori H, Yoshida S, Ashida K, Nakamura K, Takahashi T, Kunugi H. Effects of a medium-chain triglyceride-based ketogenic formula on cognitive function in patients with mild-to-moderate Alzheimer's disease. Neurosci Lett. 2019 Jan 18;690:232-236. doi: 10.1016/j.neulet.2018.10.048. Epub 2018 Oct 24. PMID 30367958
- [Background] Jensen NJ, Nilsson M, Ingerslev JS, Olsen DA, Fenger M, Svart M, Moller N, Zander M, Miskowiak KW, Rungby J. Effects of beta-hydroxybutyrate on cognition in patients with type 2 diabetes. Eur J Endocrinol. 2020 Feb;182(2):233-242. doi: 10.1530/EJE-19-0710. PMID 31821157
- [Background] Fortier M, Castellano CA, Croteau E, Langlois F, Bocti C, St-Pierre V, Vandenberghe C, Bernier M, Roy M, Descoteaux M, Whittingstall K, Lepage M, Turcotte EE, Fulop T, Cunnane SC. A ketogenic drink improves brain energy and some measures of cognition in mild cognitive impairment. Alzheimers Dement. 2019 May;15(5):625-634. doi: 10.1016/j.jalz.2018.12.017. Epub 2019 Apr 23. PMID 31027873
- [Background] Fortier M, Castellano CA, St-Pierre V, Myette-Cote E, Langlois F, Roy M, Morin MC, Bocti C, Fulop T, Godin JP, Delannoy C, Cuenoud B, Cunnane SC. A ketogenic drink improves cognition in mild cognitive impairment: Results of a 6-month RCT. Alzheimers Dement. 2021 Mar;17(3):543-552. doi: 10.1002/alz.12206. Epub 2020 Oct 26. PMID 33103819
- [Background] Cunnane S, Nugent S, Roy M, Courchesne-Loyer A, Croteau E, Tremblay S, Castellano A, Pifferi F, Bocti C, Paquet N, Begdouri H, Bentourkia M, Turcotte E, Allard M, Barberger-Gateau P, Fulop T, Rapoport SI. Brain fuel metabolism, aging, and Alzheimer's disease. Nutrition. 2011 Jan;27(1):3-20. doi: 10.1016/j.nut.2010.07.021. Epub 2010 Oct 29. PMID 21035308
- [Background] Dienel GA. Brain Glucose Metabolism: Integration of Energetics with Function. Physiol Rev. 2019 Jan 1;99(1):949-1045. doi: 10.1152/physrev.00062.2017. PMID 30565508
- [Background] Onyango IG, Dennis J, Khan SM. Mitochondrial Dysfunction in Alzheimer's Disease and the Rationale for Bioenergetics Based Therapies. Aging Dis. 2016 Mar 15;7(2):201-14. doi: 10.14336/AD.2015.1007. eCollection 2016 Mar. PMID 27114851
- [Background] Aldana BI. Microglia-Specific Metabolic Changes in Neurodegeneration. J Mol Biol. 2019 Apr 19;431(9):1830-1842. doi: 10.1016/j.jmb.2019.03.006. Epub 2019 Mar 13. PMID 30878483
- [Background] An Y, Varma VR, Varma S, Casanova R, Dammer E, Pletnikova O, Chia CW, Egan JM, Ferrucci L, Troncoso J, Levey AI, Lah J, Seyfried NT, Legido-Quigley C, O'Brien R, Thambisetty M. Evidence for brain glucose dysregulation in Alzheimer's disease. Alzheimers Dement. 2018 Mar;14(3):318-329. doi: 10.1016/j.jalz.2017.09.011. Epub 2017 Oct 19. PMID 29055815
- [Background] Myette-Cote E, Soto-Mota A, Cunnane SC. Ketones: potential to achieve brain energy rescue and sustain cognitive health during ageing. Br J Nutr. 2022 Aug 14;128(3):407-423. doi: 10.1017/S0007114521003883. Epub 2021 Sep 28. PMID 34581265
- [Background] Stagg DB, Gillingham JR, Nelson AB, Lengfeld JE, d'Avignon DA, Puchalska P, Crawford PA. Diminished ketone interconversion, hepatic TCA cycle flux, and glucose production in D-beta-hydroxybutyrate dehydrogenase hepatocyte-deficient mice. Mol Metab. 2021 Nov;53:101269. doi: 10.1016/j.molmet.2021.101269. Epub 2021 Jun 8. PMID 34116232
- [Background] Falkenhain K, Daraei A, Forbes SC, Little JP. Effects of Exogenous Ketone Supplementation on Blood Glucose: A Systematic Review and Meta-analysis. Adv Nutr. 2022 Oct 2;13(5):1697-1714. doi: 10.1093/advances/nmac036. PMID 35380602
- [Background] Newman JC, Verdin E. beta-Hydroxybutyrate: A Signaling Metabolite. Annu Rev Nutr. 2017 Aug 21;37:51-76. doi: 10.1146/annurev-nutr-071816-064916. PMID 28826372
- [Background] Myette-Cote E, Caldwell HG, Ainslie PN, Clarke K, Little JP. A ketone monoester drink reduces the glycemic response to an oral glucose challenge in individuals with obesity: a randomized trial. Am J Clin Nutr. 2019 Dec 1;110(6):1491-1501. doi: 10.1093/ajcn/nqz232. PMID 31599919
- [Background] Lowder J, Fallah S, Venditti C, Musa-Veloso K, Kotlov V. An open-label, acute clinical trial in adults to assess ketone levels, gastrointestinal tolerability, and sleepiness following consumption of (R)-1,3-butanediol (Avela). Front Physiol. 2023 Jun 28;14:1195702. doi: 10.3389/fphys.2023.1195702. eCollection 2023. PMID 37457035
- [Background] Mah E, Blonquist TM, Kaden VN, Beckman D, Boileau AC, Anthony JC, Stubbs BJ. A randomized, open-label, parallel pilot study investigating metabolic product kinetics of the novel ketone ester, bis-hexanoyl (R)-1,3-butanediol, over one week of ingestion in healthy adults. Front Physiol. 2023 Jun 22;14:1196535. doi: 10.3389/fphys.2023.1196535. eCollection 2023. PMID 37427402
- [Background] Bolyard ML, Graziano CM, Fontaine KR, Sayer RD, Fisher G, Plaisance EP. Tolerability and Acceptability of an Exogenous Ketone Monoester and Ketone Monoester/Salt Formulation in Humans. Nutrients. 2023 Nov 22;15(23):4876. doi: 10.3390/nu15234876. PMID 38068734
- [Background] Stubbs BJ, Cox PJ, Kirk T, Evans RD, Clarke K. Gastrointestinal Effects of Exogenous Ketone Drinks are Infrequent, Mild, and Vary According to Ketone Compound and Dose. Int J Sport Nutr Exerc Metab. 2019 Nov 1;29(6):596-603. doi: 10.1123/ijsnem.2019-0014. PMID 31034254
- [Background] McNelly A, Langan A, Bear DE, Page A, Martin T, Seidu F, Santos F, Rooney K, Liang K, Heales SJ, Baldwin T, Alldritt I, Crossland H, Atherton PJ, Wilkinson D, Montgomery H, Prowle J, Pearse R, Eaton S, Puthucheary ZA. A pilot study of alternative substrates in the critically Ill subject using a ketogenic feed. Nat Commun. 2023 Dec 15;14(1):8345. doi: 10.1038/s41467-023-42659-8. PMID 38102152
- [Background] Mikkelsen KH, Seifert T, Secher NH, Grondal T, van Hall G. Systemic, cerebral and skeletal muscle ketone body and energy metabolism during acute hyper-D-beta-hydroxybutyratemia in post-absorptive healthy males. J Clin Endocrinol Metab. 2015 Feb;100(2):636-43. doi: 10.1210/jc.2014-2608. Epub 2014 Nov 21. PMID 25415176
- [Background] Cunnane SC, Courchesne-Loyer A, St-Pierre V, Vandenberghe C, Pierotti T, Fortier M, Croteau E, Castellano CA. Can ketones compensate for deteriorating brain glucose uptake during aging? Implications for the risk and treatment of Alzheimer's disease. Ann N Y Acad Sci. 2016 Mar;1367(1):12-20. doi: 10.1111/nyas.12999. Epub 2016 Jan 14. PMID 26766547
- [Background] Courchesne-Loyer A, Croteau E, Castellano CA, St-Pierre V, Hennebelle M, Cunnane SC. Inverse relationship between brain glucose and ketone metabolism in adults during short-term moderate dietary ketosis: A dual tracer quantitative positron emission tomography study. J Cereb Blood Flow Metab. 2017 Jul;37(7):2485-2493. doi: 10.1177/0271678X16669366. Epub 2016 Jan 1. PMID 27629100
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Soto-Mota A, Vansant H, Evans RD, Clarke K. Safety and tolerability of sustained exogenous ketosis using ketone monoester drinks for 28 days in healthy adults. Regul Toxicol Pharmacol. 2019 Dec;109:104506. doi: 10.1016/j.yrtph.2019.104506. Epub 2019 Oct 23. PMID 31655093
- [Background] Avgerinos KI, Mullins RJ, Egan JM, Kapogiannis D. Ketone Ester Effects on Biomarkers of Brain Metabolism and Cognitive Performance in Cognitively Intact Adults >/= 55 Years Old. A Study Protocol for a Double-Blinded Randomized Controlled Clinical Trial. J Prev Alzheimers Dis. 2022;9(1):54-66. doi: 10.14283/jpad.2022.3. PMID 35098974
- [Background] Kapogiannis D, Avgerinos KI. Brain glucose and ketone utilization in brain aging and neurodegenerative diseases. Int Rev Neurobiol. 2020;154:79-110. doi: 10.1016/bs.irn.2020.03.015. Epub 2020 Jul 10. PMID 32739015
- [Background] Hohn S, Dozieres-Puyravel B, Auvin S. History of dietary treatment from Wilder's hypothesis to the first open studies in the 1920s. Epilepsy Behav. 2019 Dec;101(Pt A):106588. doi: 10.1016/j.yebeh.2019.106588. Epub 2019 Oct 30. PMID 31677579
- [Background] Khan BA, Perkins AJ, Gao S, Hui SL, Campbell NL, Farber MO, Chlan LL, Boustani MA. The Confusion Assessment Method for the ICU-7 Delirium Severity Scale: A Novel Delirium Severity Instrument for Use in the ICU. Crit Care Med. 2017 May;45(5):851-857. doi: 10.1097/CCM.0000000000002368. PMID 28263192
- [Background] Clarke K, Tchabanenko K, Pawlosky R, Carter E, Todd King M, Musa-Veloso K, Ho M, Roberts A, Robertson J, Vanitallie TB, Veech RL. Kinetics, safety and tolerability of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate in healthy adult subjects. Regul Toxicol Pharmacol. 2012 Aug;63(3):401-8. doi: 10.1016/j.yrtph.2012.04.008. Epub 2012 May 3. PMID 22561291
- [Background] White H, Venkatesh B, Jones M, Kruger PS, Walsham J, Fuentes H. Inducing ketogenesis via an enteral formulation in patients with acute brain injury:a phase II study. Neurol Res. 2020 Apr;42(4):275-285. doi: 10.1080/01616412.2019.1709743. Epub 2020 Feb 26. PMID 32098578
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Cunnane SC, Courchesne-Loyer A, Vandenberghe C, St-Pierre V, Fortier M, Hennebelle M, Croteau E, Bocti C, Fulop T, Castellano CA. Can Ketones Help Rescue Brain Fuel Supply in Later Life? Implications for Cognitive Health during Aging and the Treatment of Alzheimer's Disease. Front Mol Neurosci. 2016 Jul 8;9:53. doi: 10.3389/fnmol.2016.00053. eCollection 2016. PMID 27458340
- [Background] Morris G, Puri BK, Maes M, Olive L, Berk M, Carvalho AF. The role of microglia in neuroprogressive disorders: mechanisms and possible neurotherapeutic effects of induced ketosis. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Apr 20;99:109858. doi: 10.1016/j.pnpbp.2020.109858. Epub 2020 Jan 7. PMID 31923453
- [Background] Jang J, Kim SR, Lee JE, Lee S, Son HJ, Choe W, Yoon KS, Kim SS, Yeo EJ, Kang I. Molecular Mechanisms of Neuroprotection by Ketone Bodies and Ketogenic Diet in Cerebral Ischemia and Neurodegenerative Diseases. Int J Mol Sci. 2023 Dec 21;25(1):124. doi: 10.3390/ijms25010124. PMID 38203294
- [Background] Yang H, Shan W, Zhu F, Wu J, Wang Q. Ketone Bodies in Neurological Diseases: Focus on Neuroprotection and Underlying Mechanisms. Front Neurol. 2019 Jun 12;10:585. doi: 10.3389/fneur.2019.00585. eCollection 2019. PMID 31244753
- [Background] Gomora-Garcia JC, Montiel T, Huttenrauch M, Salcido-Gomez A, Garcia-Velazquez L, Ramiro-Cortes Y, Gomora JC, Castro-Obregon S, Massieu L. Effect of the Ketone Body, D-beta-Hydroxybutyrate, on Sirtuin2-Mediated Regulation of Mitochondrial Quality Control and the Autophagy-Lysosomal Pathway. Cells. 2023 Feb 2;12(3):486. doi: 10.3390/cells12030486. PMID 36766827
- [Background] Gnorich J, Reifschneider A, Wind K, Zatcepin A, Kunte ST, Beumers P, Bartos LM, Wiedemann T, Grosch M, Xiang X, Fard MK, Ruch F, Werner G, Koehler M, Slemann L, Hummel S, Briel N, Blume T, Shi Y, Biechele G, Beyer L, Eckenweber F, Scheifele M, Bartenstein P, Albert NL, Herms J, Tahirovic S, Haass C, Capell A, Ziegler S, Brendel M. Depletion and activation of microglia impact metabolic connectivity of the mouse brain. J Neuroinflammation. 2023 Feb 24;20(1):47. doi: 10.1186/s12974-023-02735-8. PMID 36829182
- [Background] Afridi R, Kim JH, Rahman MH, Suk K. Metabolic Regulation of Glial Phenotypes: Implications in Neuron-Glia Interactions and Neurological Disorders. Front Cell Neurosci. 2020 Feb 11;14:20. doi: 10.3389/fncel.2020.00020. eCollection 2020. PMID 32116564
- [Background] Bernier LP, York EM, Kamyabi A, Choi HB, Weilinger NL, MacVicar BA. Microglial metabolic flexibility supports immune surveillance of the brain parenchyma. Nat Commun. 2020 Mar 25;11(1):1559. doi: 10.1038/s41467-020-15267-z. PMID 32214088
- [Background] Cunnane SC, Trushina E, Morland C, Prigione A, Casadesus G, Andrews ZB, Beal MF, Bergersen LH, Brinton RD, de la Monte S, Eckert A, Harvey J, Jeggo R, Jhamandas JH, Kann O, la Cour CM, Martin WF, Mithieux G, Moreira PI, Murphy MP, Nave KA, Nuriel T, Oliet SHR, Saudou F, Mattson MP, Swerdlow RH, Millan MJ. Brain energy rescue: an emerging therapeutic concept for neurodegenerative disorders of ageing. Nat Rev Drug Discov. 2020 Sep;19(9):609-633. doi: 10.1038/s41573-020-0072-x. Epub 2020 Jul 24. PMID 32709961
- [Background] Fu C, Weng S, Liu D, Guo R, Chen M, Shi B, Weng J. Review on the Role of Mitochondrial Dysfunction in Septic Encephalopathy. Cell Biochem Biophys. 2025 Mar;83(1):135-145. doi: 10.1007/s12013-024-01493-5. Epub 2024 Aug 30. PMID 39212823
- [Background] Preau S, Vodovar D, Jung B, Lancel S, Zafrani L, Flatres A, Oualha M, Voiriot G, Jouan Y, Joffre J, Uhel F, De Prost N, Silva S, Azabou E, Radermacher P. Energetic dysfunction in sepsis: a narrative review. Ann Intensive Care. 2021 Jul 3;11(1):104. doi: 10.1186/s13613-021-00893-7. PMID 34216304
- [Background] Zhang J, Chen S, Hu X, Huang L, Loh P, Yuan X, Liu Z, Lian J, Geng L, Chen Z, Guo Y, Chen B. The role of the peripheral system dysfunction in the pathogenesis of sepsis-associated encephalopathy. Front Microbiol. 2024 Jan 17;15:1337994. doi: 10.3389/fmicb.2024.1337994. eCollection 2024. PMID 38298892
- [Background] Kealy J, Murray C, Griffin EW, Lopez-Rodriguez AB, Healy D, Tortorelli LS, Lowry JP, Watne LO, Cunningham C. Acute Inflammation Alters Brain Energy Metabolism in Mice and Humans: Role in Suppressed Spontaneous Activity, Impaired Cognition, and Delirium. J Neurosci. 2020 Jul 15;40(29):5681-5696. doi: 10.1523/JNEUROSCI.2876-19.2020. Epub 2020 Jun 8. PMID 32513828
- [Background] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265